CLINICAL TRIAL: NCT04074863
Title: Norwegian Distal Ulna Resection vs. Replacement Study. A Prospective Randomized Multicenter Study
Brief Title: Norwegian Distal Ulna Resection - Replacement Study
Acronym: NORDURR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Istvan Zoltan Rigo, Consultant, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OstfoldHT
Record Dates: First submitted 2019-03-28; First posted 2019-08-30 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis Wrist
Keywords: Distal radioulnar joint; Darrach procedure; Ulnar head resection; Herbert prosthesis; Ulnar head replacement
MeSH Terms: interventions — Prostheses and Implants

STUDY DESIGN:
Intervention Model Description: Participants randomized to one of the group and receive the group specific surgery. Postoperative treatment is identical between the groups.
Who Masked: Outcomes Assessor
Masking Description: An independent hand therapist, who is not involved in the rehabilitation of the participants, will carry out the measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Darrach (Active Comparator): Surgical procedure: resection of distal ulna
  Interventions: Procedure: Darrach
- Prosthesis (Active Comparator): Surgical procedure: ulnar head replacement
  Interventions: Procedure: Prosthesis

INTERVENTIONS:
Procedure: Darrach — Surgical treatment of painful DRU osteoarthritis with resection of distal ulna
  Other Names: resection of ulnar head (Darrach procedure)
  Arms: Darrach
Procedure: Prosthesis — Surgical treatment of painful DRU osteoarthritis with distal ulna replacement with Herbert implant
  Other Names: Herbert disltal ulna implant
  Arms: Prosthesis

SUMMARY:
Osteoarthritis of the joint between the forearm bones at the wrist (distal radioulnar joint, DRUJ) is a common sequel of fracture and ligament injuries or degenerative disease of the wrist. Intact DRUJ is important for normal load transfer from the hand to the forearm. DRUJ osteoarthritis leads to pain and decreased lifting capacity and rotation of the forearm. The standard treatment is resection of the ulnar head, known as the Darrach procedure. After the resection there is no longer contact in the affected joint, however, some patients can experience instability or impingement between the forearm bones. With ulnar head implant replacement may the load transfer and the stability between the forearm bones less affected. Studies with good long term results are published with both resection and replacement. However, these methods were never compared and thus it is not clear, which of the methods gives the best clinical result and less complications.

The aim of this study is to compare Darrach procedure with ulnar head replacement in a prospective randomized multicenter study. Several hand surgical centers form Norway would participate this study.

Individuals seeking treatment for their stable but painful DRUJ joints will be included and randomized to either Darrach procedure or ulnar head implant. Participants will be followed up to 5 years. Range of motion and grip strength measures and functional scores would be registered before operation, after 3 months, 1 and 5 years. Eventual complications and reoperations would be also registered.

DETAILED DESCRIPTION:
Osteoarthritis of the joint between the forearm bones at the wrist (distal radioulnar joint, DRUJ) is a common sequel of fracture and ligament injuries or degenerative disease of the wrist. Intact DRUJ is important for normal load transfer from the hand to the forearm. DRUJ osteoarthritis leads to pain and decreased lifting capacity and rotation of the forearm. The standard treatment is resection of the ulnar head, known as the Darrach procedure. After the resection there is no longer contact in the affected joint, however, some patients can experience instability or impingement between the forearm bones. With ulnar head implant replacement may the load transfer and the stability between the forearm bones less affected. Studies with good long term results are published with both resection and replacement. However, these methods were never compared and thus it is not clear, which of the methods gives the best clinical result and less complications.

The aim of this study is to compare Darrach procedure with ulnar head replacement in a prospective randomized multicenter study. The study would be coordinated from Østfold Hospital Trust, and Oslo University Hospital, Haukeland University Hospital, Innlandet Hospital Trust, University Hospital of St Olav and University Hospital of North Norway would participate this study.

Participants would be included among individuals seeking treatment for their stable but painful DRUJ joints. Informed consent will be gained from every participant. The group size was calculated to 20 participants in both groups.

Participants will be randomized to either Darrach procedure or ulnar head implant. The procedures would be carried out standardized in every center. No further stabilization procedure for the ulna stump would be used in resection. Herbert UHP implant (Herbert Ulnar Head Prosthesis, KLS Martin, Germany) would be used for ulnar head replacement. Postoperative treatment and follow up would be identical between the groups.

Range of motion and grip strength measures and functional scores would be registered by an independent hand therapist before operation, after 3 months, 1 and 5 years. Eventual complications and reoperations would be also registered.

Patient related outcome measure scores, range of motion and grip strength would be registered as outcomes. The results would be checked for normal distribution and either parametric or non parametric statistical tests would be chosen for comparison of the two groups.

The null hypothesis is that Darrach procedure and ulnar head replacement with implant gives similar functional results, similar frequency of complication and reoperations.

ELIGIBILITY:
Inclusion Criteria:

* painful osteoarthritis distal radioulnar joint
* stable DRUJ

Exclusion Criteria:

* activ inflammatory disease with significant destruction of the joint
* "low demand" persons
* significant instability i DRUJ
* active infections, poor soft tissue conditions
* accidental wound on the operated hand
* general contraindications for surgery

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Norwegian version of Quick DASH (Quick Disability Arm Shoulder Hand) score | at 5 years
  specific patient reported outcome measure, scale with range 0-100, with 0 defined as best possible and 100 as worst possible outcome

SECONDARY OUTCOMES:
Norwegian vesrion of PRWHE (Patient Rated Wrist Hand Evaluation) score | at 5 years
  Hand specific patient reported outcome measure, scale with range 0-100, with 0 defined as best and 100 as worst subjective outcome
Visual Analogue Scale (VAS) pain scale | at 5 years
  subjective evaluation of pain intensity, a scale with range 0-10 with 0 defined as best possible and 10 as worst outcome
Active range of motion | at 5 years
  objective measurement of movements in degrees, a scale with range 0-180 degrees.
Grip strength | at 5 years
  Measurement of grip strength of the hand, scale with range 0-100 kilograms
complications and reoperations | at 5 years
  Registration of occurance of any adverse event, will be reported as number of participants with complications and reoperations

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Zoltan Rigo, PhD, Principal Investigator — Ostfold Hospital Trust
Locations (6):
- Norway (6):
  - Innlandet Hospital Trust, Lillehammer, Oppland
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - University Hospital of St Olav, Trondheim
  - Østfold Hospital Trust, Moss, Østfold fylke

IPD SHARING:
Plan to Share IPD: No